CLINICAL TRIAL: NCT04604613
Title: Prediction of Recurrence Among Low Risk Endometrial Cancer Population
Brief Title: Prediction of Recurrence Among Low Risk Endometrial Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA12-0550; NCI-2020-07548 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA12-0550 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: FIGO Grade 1 Endometrial Endometrioid Adenocarcinoma; FIGO Grade 2 Endometrial Endometrioid Adenocarcinoma
MeSH Terms: interventions — Ovariectomy; Hysterectomy; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biospecimen collection, node mapping): Patients undergo hysterectomy and sentinel lymph node mapping. Patients may also undergo bilateral salpingo-oophorectomy at the direction of the treating physician. If peritoneal disease or other contraindications to lymphatic mapping are detected at the time of surgery, mapping and sentinel node biopsy are performed at the surgeon's discretion. At the time of hysterectomy, patients undergo collection of tissue for molecular testing. Before and after surgery, patients also undergo collection of blood samples for tumor marker analysis.
  Interventions: Procedure: Bilateral Salpingectomy with Oophorectomy; Procedure: Biospecimen Collection; Procedure: Hysterectomy; Other: Laboratory Biomarker Analysis; Procedure: Lymph Node Mapping; Procedure: Sentinel Lymph Node Biopsy

INTERVENTIONS:
Procedure: Bilateral Salpingectomy with Oophorectomy — Undergo standard of care bilateral salpingo-oophorectomy
  Other Names: bilateral salpingo-oophorectomy
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples
Procedure: Hysterectomy — Undergo standard of care hysterectomy
  Other Names: Hysterectomy NOS
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Lymph Node Mapping — Undergo sentinel lymph node mapping
  Other Names: lymphatic mapping
Procedure: Sentinel Lymph Node Biopsy — Undergo sentinel lymph node biopsy
  Other Names: Sentinel Node Biopsy; Sentinel node biopsy alone; SLNB; SNB

SUMMARY:
This study investigates whether molecular testing can help to predict the risk of endometrial cancer coming back (recurrence) after treatment in patients diagnosed with low risk endometrial cancer and scheduled to have surgery to remove the uterus and/or cervix (hysterectomy). Having sentinel lymph node mapping performed may help researchers to see if the cancer has spread in patients with low risk endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Validate the use of a molecular panel of estrogen-induced genes to predict recurrence in low risk endometrial cancer.

SECONDARY OBJECTIVES:

I. Calculate the positive predictive value (PPV)/negative predictive value (NPV)/sensitivity (Sens)/specificity (Spec) of lymph node mapping to predict pelvic lymph node involvement.

II. Correlate CA125 and HE4 levels with recurrence and to explore the use of other serum biomarkers to predict recurrence.

III. Describe patterns of recurrence in a low risk patient population. IV. Determine if molecular panel can predict lymph node involvement in low risk endometrial cancer patients who undergo pelvic and para-aortic lymphadenectomy.

V. Compare performance of molecular panel to the Mayo low risk criteria for prediction of lymph node involvement.

VI. Compare performance of molecular panel to the high intermediate risk criteria from Gynecologic Oncology Group, trial 99 (GOG 99) for prediction of recurrence.

VII. Determine the feasibility of lymph node mapping in this patient population.

VIII. Determine the morbidity and mortality of lymph node dissection and mapping.

OUTLINE:

Patients undergo hysterectomy and sentinel lymph node mapping. Patients may also undergo bilateral salpingo-oophorectomy at the direction of the treating physician. If peritoneal disease or other contraindications to lymphatic mapping are detected at the time of surgery, mapping and sentinel node biopsy are performed at the surgeon's discretion. At the time of hysterectomy, patients undergo collection of tissue for molecular testing. Before and after surgery, patients also undergo collection of blood samples for tumor marker analysis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed low grade (grade 1-2) endometrioid type adenocarcinoma
* Candidate for surgery
* No evidence of deep invasion or peritoneal disease in patients that have undergone preoperative imaging
* Patients may have had prior hormonal treatment for the treatment of early endometrial neoplasia. Patients may not have had prior radiation or chemotherapy for treatment of endometrial cancer
* Patients must have a negative pregnancy if of childbearing potential

Exclusion Criteria:

* Histologically confirmed high grade endometrioid or non-endometrioid type endometrial cancer (including serous, clear cell, carcinosarcoma or any mixed tumor containing these cell types)
* Medical co-morbidities making surgery unsafe, as determined by the primary treating physician
* Evidence of deep myometrial invasion, cervical involvement or peritoneal disease on preoperative imaging
* Prior treatment with radiation or chemotherapy for endometrial cancer
* Any contraindication to lymph node mapping

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with low risk endometrial cancer who are scheduled to have a hysterectomy
Sampling Method: Non-Probability Sample
Enrollment: 518 (Actual)
Dates: Start 2012-11-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence | At 2 years
  Will validate a model's ability to predict 2-year recurrence in low-risk endometrial cancer patients.

SECONDARY OUTCOMES:
Predictive ability of lymph node mapping in pelvic lymph node involvement | Up to 2 years
  Will calculate the sensitivity (true positive fraction [TPF]), specificity (1-false positive fraction [FPF]), positive predictive value (PPV), and negative predictive value (NPV) of lymph node mapping in predicting pelvic lymph node involvement, along with 2-sided 95% confidence intervals.
Feasibility of lymph node mapping | Up to 2 years
  Feasibility of lymph node mapping in this patient population will be determined after examining the TPF, FPF, PPV, and NPV.
Morbidity and mortality prevalence associated with lymph node dissection | Up to 2 years
  Morbidity and mortality prevalence associated with lymph node dissection and mapping will be calculated with 95% confidence intervals.
Patterns of recurrence | Up to 2 years
  Will determine which demographic and clinical traits are most associated with recurrence rate using proportional hazards models and with 2-year recurrence using logistic regression models. Will conduct univariate analyses using log-rank tests and Fisher's exact tests, in the case of categorical traits, and proportional hazards and logistic regression models, in the case of continuous traits. Will examine all traits for violations of the proportional hazards assumption (recurrence rate models), and will examine all continuous traits for functional form (recurrence and recurrence rate models). Will use the same methods to determine whether CA125 and HE4 is associated with recurrence and recurrence rate.
Predictive ability of molecular panel in lymph node involvement | Up to 2 years
  Will use Cartesian and Regression Tree Analysis and logistic regression to determine if the molecular panel can predict lymph node involvement. Will assess the use of the model by calculating sensitivity, specificity, PPV, and NPV. Additionally, will examine how often the results of the molecular panel model concur with the Mayo low risk criteria for prediction of lymph node involvement. All agreement statistics will be presented with their 95% confidence intervals.
Predictive ability of marker panel in recurrence | Up to 2 years
  Will examine how well the predictive ability of the marker panel agrees with the predictive ability of the high intermediate risk criteria from Gynecologic Oncology Group, trial 99 using this patient population. 95% confidence intervals will be calculated for all concordance statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon N Westin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org